CLINICAL TRIAL: NCT04451785
Title: Relationships Between Hemolysis, Erythrosis, Circulating Microparticles and Vascular Function in Patients With Hereditary Spherocytosis
Brief Title: Hereditary Spherocytosis and Vascular Function
Acronym: VASCUSPHERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0949; 2019-A03203-54 (Other: ID-RCB)
Record Dates: First submitted 2020-06-18; First posted 2020-06-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2024-04

CONDITIONS: Hereditary Spherocytosis
Keywords: Hereditary spherocytosis; hemolysis; microparticles; vascular function; red blood cell
MeSH Terms: conditions — Spherocytosis, Hereditary; Hemolysis | interventions — Blood Specimen Collection; Pulse Wave Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy individuals (Active Comparator): 20 healthy subjets aged 6 years minimum will be included in this study. This is the control group.
  Interventions: Biological: blood sample; Diagnostic Test: Pulse wave velocity
- Patients with hereditary spherocytosis (Experimental): 60 patients with hereditary spherocytosis will be included in this study.
  Interventions: Biological: blood sample; Diagnostic Test: Pulse wave velocity

INTERVENTIONS:
Biological: blood sample — 6 tubes of 4 milliliters (ml) maximum (total: 24 ml) will be sampled for the measurements of the different biological markers. In case of the genetic mutation is already known, only 5 tubes will be collected (total: 20 ml).
Diagnostic Test: Pulse wave velocity — Non-invasive measurement of pulse wave velocity between the carotid and femoral arteries with piezo-electric sensors.

SUMMARY:
Background : Patients with hereditary spherocytosis (HS) are characterized by increased red blood cell (RBC) fragility and a loss of RBC deformability. While the clinical variability of the disease may be heterogenous from one patient to another, some studies reported the occurrence of vascular complications, notably in patients who have been splenectomized.

Purpose : The aim of the study is to test the associations between the degree of vascular dysfunction and the extent of hemolysis, the amount of circulating microparticles, the level of erythrosis and the degree of RBC biophysical alterations.

Abstract : Recent studies reported the occurrence of vascular complications in patients with HS, notably in patients who have previously been splenectomized. However, the exact reasons of these complications are unknown and no study investigated the vascular function in HS patients.

Main objective Highlight the presence of altered vascular function in HS patients and test the relationships with the level of hemolysis and circulating microparticles.

Secondary objectives To evaluate the associations between clinical severity and 1) the level of vascular dysfunction and 2) several biomarkers (hemolysis, hematological parameters, circulating microparticles, erythrosis, RBC biophysical properties).

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

* age ≥ 6 years old
* written, informed and signed consent by the healthy volunteer, or by both parents or legal guardian if the healthy volunteer is a minor
* Healthy volunteer affiliated to a social security scheme or assimilated
* Healthy volunteer not subject to any legal protection measure

Patients with hereditary spherocytosis:

* age ≥ 6 years old
* Patient with hereditary or non-splenectomized spherocytosis
* Written, informed and signed consent by the patient, or by at least one of the two parents or legal guardian if the patient is a minor
* Patient affiliated to a social security scheme or assimilated
* Patient not subject to any legal protection measure

Exclusion Criteria:

Healthy controls:

* Pregnant or lactating woman
* Subjects with hereditary spherocytosis or other characterized condition by chronic hemolysis
* Subjects with known pathology affecting the vascular system
* Blood donation (less than a month old)
* Not affiliated to a social security scheme
* Patient participating in another interventional research protocol that may interfere with this protocol (according to the investigator's judgment).

Patients with hereditary spherocytosis:

* Patient who received a blood transfusion in the 3 months preceding
* Pregnant or lactating woman
* Any disease or condition other than hereditary spherocytosis, chronic or not, likely to induce chronic or acute intravascular hemolysis
* Patient participating in another interventional research protocol that may interfere with this protocol (according to the investigator's judgment).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
measurement of pulse wave velocity (PWV) | Day 1
  Vascular function (arterial stiffness) will be investigated by the measurement of pulse wave velocity (PWV). Vascular dysfunction will be defined by a PWV value higher than 6 meter/second (m/s) and 10 m/s in children and adults with HS, respectively.

SECONDARY OUTCOMES:
Hemogram | Day 1
  The hemogram is a complete blood count of the different cell types. All these measures are performed simultaneously on a standard hematology analyzer.
Markers of hemolysis | Day 1
  These markers are measured simultaneously on a standard biochemistry analyzer
Circulating microparticles | Day 1
  Circulating microparticles of various cell origin will be measured by flow cytometry
Markers of erythrosis | Day 1
  Markers of erythrosis (i.e., suicidal death of red blood cells) will be measured by flow cytometry
Blood viscosity | Day 1
  Blood viscosity (expressed in Pa.s) will be measured on a cone-plate viscosimeter, ektacytometry and light transmission, respectively.
Red blood cell deformability | Day 1
  Red blood cell deformability will be measured simultaneously on a Lorrca ektacytometry (Laser-assisted Rotational Red Cell Analyser).
Red blood cell aggregation | Day 1
  Red blood cell aggregation will be measured simultaneously on a Lorrca ektacytometry (Laser-assisted Rotational Red Cell Analyser).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut d'Hématologie et Oncologie PEdiatrique (iHOPe), Lyon
  - Hôpital Edouard Herriot, Lyon

REFERENCES:
- [Result] Casabianca M, Gauthier A, Nader E, Cannas G, Martin F, Martin M, Carin R, Boisson C, Guillot N, Merazga S, Renoux C, Bertrand Y, Garnier N, Hot A, Muniansi I, Halfon-Domenech C, Poutrel S, Joly P, Connes P. Red blood cell senescence and vascular function in patients with hereditary spherocytosis with and without splenectomy. Br J Haematol. 2024 May;204(5):e41-e44. doi: 10.1111/bjh.19444. Epub 2024 Apr 2. No abstract available. PMID 38563320